CLINICAL TRIAL: NCT03686579
Title: Chest Trauma:Prediction of Associated Thoracic Injuries by Clinical and Radiological Studies .Specificity and Sensitivity
Brief Title: Chest Trauma :Prediction of Thoracic Injuries Clinically and Radiologically
Acronym: chesttrauma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, alzahraa gamal hasanein, Chest trauma: prediction of associated thoracic injuries by clinical and radiological studies .specificity and sensitivity, Assiut University
Other Study IDs: CT
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Chest Trauma; Fluid Balance; Disorder
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chest trauma: 1. Early detection and diagnosis of associated thoracic injuries .
  2. decrease of costs required for investigations . 3- sensitivity and specificity of the investigations
  Interventions: Radiation: chest trauma

INTERVENTIONS:
Radiation: chest trauma — clinical and radiological study

SUMMARY:
• Trauma is a major cause of morbidity and mortality worldwide. Despite the advent of specialized trauma centers the outcome of patients who sustain major trauma remains disappointing. Plain radiography and more advanced imaging techniques such as ultrasound, computerised tomography (CT) and angiography, have a major role to play in the early decision making and subsequent management of patients who sustain polytrauma. This article discusses the choice of emergency imaging techniques available in chest trauma for clinicians and radiologists; their evaluation and some of the common pitfalls that may lead to errors of interpretation.

DETAILED DESCRIPTION:
Imaging plays a key role for both, the primary diagnostic work-up, and the secondary assessment of potential treatment. Despite its well-known limitations, the posteroanterior chest radiograph remains the starting point of the imaging work-up. Adjunctive imaging with computed tomography, that recently is increasingly often performed on multidetector computed tomography units, adds essential information not readily available on the conventional radiograph. This allows better definition of trauma-associated thoracic injuries not only in acute traumatic aortic injury, but also in pulmonary, tracheobronchial, cardiac, diaphragmal, and thoracic skeletal injuries. This article reviews common radiographic findings in patients after chest trauma, shows typical imaging features resulting from thoracic injury, presents imaging algorithms, and recalls to the reader less common but clinically relevant entities encountered in patients after thoracic trauma.

ELIGIBILITY:
Inclusion Criteria:

* chest trauma 2. recent trauma: presented within48 h

Exclusion Criteria:

* Old trauma more than 48h 2-Pt transferred urgently to operating room

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Information collected by this study may contribute to the care of patients in the future who have the same lesions as those that participate in this study. The information may also improve the future management of study participants. On the other hand patients will benefit from the clinical and radiological follow up postoperatively. There are no known risks associated with participation in this study. Patients' treatment and follow up will not be altered by any means
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
detection of associated thoracic injuries : fracture rib ,sternum…. etc detection of sensitivity and specificity of clinical and radiological finding detection of associated thoracic injuries : fracture rib ,sternum…. etc | after one week
  prediction of associated thoracic injuries by clinical and radiological studies .specificity and sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Alzahraa gamal hasanien sayed, Principal Investigator — Assiut University